CLINICAL TRIAL: NCT01028651
Title: An Open-Label Study to Assess the Safety and Efficacy of Treprostinil to Facilitate Liver Transplantation in Patients With Portopulmonary Hypertension
Brief Title: A Study to Assess the Safety and Efficacy of Treprostinil to Facilitate Liver Transplantation in Patients With Portopulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: United Therapeutics (Industry)
Collaborators: University of California, Los Angeles (Other); Brigham and Women's Hospital (Other); University of Texas (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: RIV-PH-414
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Portopulmonary Hypertension; Pulmonary Arterial Hypertension; Pulmonary Hypertension
Keywords: PAH; Pulmonary Hypertension; Remodulin; Treprostinil; Quality of Life
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Portopulmonary hypertension
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — Remodulin is supplied in concentrations of 1, 2.5 , 5, and 10 mg/mL and can be administered as supplied or diluted for intravenous (IV) infusion prior to administration.
  Remodulin is indicated for subcutaneous (SC) or IV use only as a continuous infusion. Remodulin is preferably infused subcutaneously, but can be administered by a central IV line if the SC route is not tolerated. The infusion rate is initiated at 1.25 ng/kg/min. If this initial dose cannot be tolerated because of systemic effects, the infusion rate should be reduced to 0.625 ng/kg/min.
  Other Names: Remodulin

SUMMARY:
This was a multicenter, prospective, observational, open-label study. Patients meeting inclusion/exclusion criteria received treatment with treprostinil as recommended by their treating physicians and were followed according to standard of care. This observational study collected clinical data and biologic specimens from patients who were treated for portopulmonary hypertension (PoPH), with a goal of achieving hemodynamic parameters appropriate for orthotopic liver transplantation candidacy, including mean pulmonary arterial pressure (mPAP) less than 35 mmHg and pulmonary vascular resistance (PVR) less than 3 Wood-units (WU) at Week 24 in patients with severe PoPH.

DETAILED DESCRIPTION:
Treprostinil is approved as a continuous subcutaneous (SC) or intravenous (IV) infusion by the FDA for the treatment of WHO group I PAH with New York Heart Association (NYHA) Functional Class II, III or IV symptomatology. To date, treprostinil has not been studied in the setting of PoPH; however, it is commonly prescribed in this setting. This was an observational, open-label, multicenter study which documented the safety and efficacy profile of this agent in PoPH to facilitate orthotopic liver transplantation (OLT).

ELIGIBILITY:
Inclusion Criteria:

* Patients must:

  1. Had portal hypertension.
  2. Be otherwise suitable candidates for OLT.
  3. Had severe pulmonary arterial hypertension (PAH) defined as a resting mean pulmonary arterial pressure (mPAP) >35 mmHg and pulmonary vascular resistance (PVR) ≥3 Wood Units (WU) by right heart catheterization (RHC) performed as part of standard of care evaluation within 90 days of enrollment.
  4. Treprostinil therapy must be recommended by the treating physician per standard of care.
  5. Be NYHA Functional Class II, III, or IV.
  6. Had pulmonary capillary wedge (PCW) pressure ≤18 mmHg and transpulmonary gradient (TPG) ≥15 mmHg.

Exclusion Criteria:

* Patients must not:

  1. Had received any any investigational therapy as part of a clinical trial for any indication within 30 days prior to enrollment.
  2. Had a change in dose of treatment for PAH (bosentan [Tracleer], ambrisentan [Letairis], tadalafil [Adcirca], or sildenafil [Revatio]), within 30 days prior to enrollment. That is, subjects may have been treated with any of these agents provided the dose was stable for at least 30 days prior to enrollment.
  3. Had renal failure requiring hemodialysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects were recruited from 4 liver transplantation centers in the US, referred for portopulmonary hypertension.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Study Director — University of California, Los Angeles; Micah Fisher, MD, Study Director — Emory University; Aaron Waxman, MD, PhD, Study Director — Brigham and Women's Hospital; Sonja Bartolome, MD, Study Director — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - Emory Univeristy, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Texas, Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Treprostinil Injection: Subjects meeting inclusion/exclusion criteria with portopulmonary hypertension (PoPH) and severe pulmonary arterial hypertension (PAH).
Period: Overall Study
Arm/Group | Treprostinil Injection
Started | 13
Completed | 10
Not Completed | 3
Not completed — Death | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (8.00)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Hemodynamic Parameters Appropriate for Orthotopic Liver Transplantation Candidacy at Week 24.
Description: The primary efficacy endpoint was the number of subjects who achieved a mean pulmonary arterial pressure (mPAP) less than 35 mmHg and a pulmonary vascular resistance (PVR) less than 3 Wood units (WU) at Week 24 in patients with severe portopulmonary hypertension (PoPH).
Time Frame: 24 Weeks
Population: The total number of subjects enrolled and analyzed.
Measure: Number; unit: participants
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
participants
  Primary endpoint achieved | 1
  Primary endpoint not achieved | 12

2. Secondary Outcome: Change in Hemodynamic Parameters (Via Right Heart Catheterization [RHC]) at Rest From Baseline to Week 24
Description: The change in hemodynamic parameters (including systolic pulmonary arterial pressure [PAPs], diastolic pulmonary arterial pressure [PAPd], mean pulmonary arterial pressure [mPAP], and transpulmonary gradient [TPG]) was evaluated at rest from Baseline to Week 24. The median change in hemodynamic parameters from Baseline to Week 24 via right-heart catheterization (RHC) is presented.
Time Frame: 24 weeks
Population: All subjects with data available at Baseline and Week 24
Measure: Median (Full Range); unit: mmHg
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
mmHg
  Mean pulmonary arterial pressure (mmHg) | -3.8 [-26 to 1]
  Systolic pulmonary arterial pressure (mmHg) | -2.0 [-46 to 1]
  Diastolic pulmonary arterial pressure (mmHg) | -4.0 [-22 to 1]
  Mean right arterial pressure (mmHg) | -2.0 [-9 to 5]
  Mean systemic arterial pressure (mmHg) | -0.7 [-28 to 34.7]
  Systolic systemic arterial pressure (mmHg) | 7.0 [-44 to 94]
  Diastolic systemic arterial pressure | 0 [-20 to 35]
  Mean pulmonary capillary wedge pressure (mmHg) | 0 [-3 to 8]
  Transpulmonary gradient (mmHg) | -6.8 [-24 to 4]

3. Secondary Outcome: Change in Heart Rate at Rest From Baseline to Week 24
Description: The change in heart rate was evaluated at rest from Baseline to Week 24.
Time Frame: 24 weeks
Population: All subjects with data available at Baseline and Week 24
Measure: Median (Full Range); unit: beats/min
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
beats/min | 0.5 [-10 to 8]

4. Secondary Outcome: Change in Cardiac Output at Rest From Baseline to Week 24
Description: The change in cardiac output was evaluated at rest from Baseline to Week 24. The median change in cardiac output from Baseline to Week 24 is presented.
Time Frame: 24 weeks
Population: All subjects with data available at Baseline and Week 24
Measure: Median (Full Range); unit: L/min
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
L/min | 0.3 [-6.5 to 4]

5. Secondary Outcome: Change in Arterial and Venous Oxygen Saturation at Rest From Baseline to Week 24
Description: The change in arterial and venous oxygen saturation was evaluated at rest from Baseline to Week 24.
Time Frame: 24 weeks
Population: All subjects with data available at Baseline and Week 24
Measure: Median (Full Range); unit: percentage bound to hemoglobin
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
percentage bound to hemoglobin
  Mixed venous oxygen saturation (%) | -2.0 [-7 to 14]
  Arterial oxygen saturation (%) | 0.5 [-2 to 2]

6. Secondary Outcome: Change in Pulmonary Vascular Resistance (PVR) at Rest From Baseline to Week 24
Description: The change in pulmonary vascular resistance (PVR) was evaluated at rest from Baseline to Week 24.
Time Frame: 24 weeks
Population: All subjects with data available at Baseline and Week 24
Measure: Median (Full Range); unit: Wood Units
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 13
Wood Units | -0.3 [-8.2 to 1.3]

7. Secondary Outcome: Change in 6-minute Walk Distance (6MWD) From Baseline to Weeks 12 and 24.
Description: The 6-Minute Walk Test was conducted at Screening, Baseline prior to starting study drug and at least 24 hours after the Screening test, and during the Treatment Phase at Weeks 12 and 24.
Time Frame: Baseline and Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24
Measure: Median (Full Range); unit: Meters
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 11
Meters
  Change from Baseline to Week 12 | 54.5 [-48 to 133]
  Change from Baseline to Week 24 | 12.0 [-18 to 90]

8. Secondary Outcome: Change in Echocardiogram Parameters (Right Atrium and Right Ventricle Area) From Baseline to Weeks 12 and 24
Description: Standard transthoracic echocardiogram with continuous wave Doppler and color flow imaging was completed at Screening. All patients who were enrolled in this study underwent an echocardiogram within 30 days of enrollment as well as repeat echocardiograms on Weeks 12 and 24.
Time Frame: Baseline and Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24.
Measure: Median (Full Range); unit: cm2
Groups:
- Treprostinil Injection-Baseline to Week 12; Treprostinil Injection-Baseline to Week 24: Subjects meeting inclusion/exclusion criteria with portopulmonary hypertension (PoPH) and severe pulmonary arterial hypertension (PAH).
Arm/Group | Treprostinil Injection-Baseline to Week 12 | Treprostinil Injection-Baseline to Week 24
Number analyzed (Participants) | 8 | 7
cm2
  Right atrium area (cm2) | -0.1 [-7.7 to 3.7] | -1.7 [-12 to 10.0]
  Right ventricle area (cm2) | -1.0 [-11 to 2.2] | -7.4 [-12 to 19.0]

9. Secondary Outcome: Change in Echocardiogram Parameters (Right Ventricle Diameter) From Baseline to Weeks 12 and 24
Description: as for outcome 8
Time Frame: Baseline and Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24.
Measure: Median (Full Range); unit: mm
Arm/Group | Treprostinil Injection-Baseline to Week 12 | Treprostinil Injection-Baseline to Week 24
Number analyzed (Participants) | 8 | 7
mm | -5.0 [-45 to 2.0] | 3.0 [-10 to 3.0]

10. Secondary Outcome: Change in Echocardiogram Parameters (Right Ventricular Systolic Pressure) From Baseline to Weeks 12 and 24
Description: as for outcome 8
Time Frame: Baseline and Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Treprostinil Injection-Baseline to Week 12 | Treprostinil Injection-Baseline to Week 24
Number analyzed (Participants) | 8 | 7
mmHg | -12 [-28 to 11.0] | -5.0 [-38 to 17.0]

11. Secondary Outcome: Change in Echocardiogram Parameters (Tricuspid Annular Plane Systolic Excursion) From Baseline to Weeks 12 and 24
Description: as for outcome 8
Time Frame: Baseline and Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24.
Measure: Median (Full Range); unit: cm
Arm/Group | Treprostinil Injection-Baseline to Week 12 | Treprostinil Injection-Baseline to Week 24
Number analyzed (Participants) | 8 | 7
cm | 0.5 [-0.5 to 0.9] | 0.1 [-0.6 to 0.8]

12. Secondary Outcome: Change in Quality of Life From Baseline to Weeks 12 and 24
Description: The 36-item Short Form Survey (SF-36) is a health related quality of life instrument, which measures dimensions of physical and social roles and functioning, mental health, vitality, and pain. Items are scored on a 0 to 100 range so that the lowest scores represent the highest disability. The quality of life assessment was conducted at Baseline and Weeks 12 and 24 and the change from Baseline to Weeks 12 and 24 is presented.
Time Frame: Baseline and Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treprostinil Injection-Baseline to Week 12 | Treprostinil Injection-Baseline to Week 24
Number analyzed (Participants) | 11 | 9
units on a scale
  Physical functioning | 5.7 [-1.9 to 19.1] | 10.5 [3.8 to 21.1]
  Role-Physical | 7.9 [-2.3 to 20.2] | 9.0 [4.5 to 27.0]
  Bodily pain | 3.6 [-4.0 to 12.5] | 6.0 [-0.8 to 10.5]
  General health | 4.5 [-2.4 to 12.8] | 3.6 [-2.4 to 18.1]
  Vitality | 5.9 [-18 to 11.9] | 7.4 [-21 to 20.8]
  Social functioning | 7.5 [-5.0 to 15.0] | 0 [0 to 25.1]
  Role-Emotional | 13.9 [-24 to 24.4] | 10.4 [-10 to 17.4]
  Mental health | 2.6 [-13 to 20.9] | 0 [-5.2 to 26.2]
  Physical component summary | 9.8 [-2.4 to 14.3] | 8.2 [5.6 to 22.0]
  Mental component summary | 7.0 [-21 to 17.8] | 2.6 [-13 to 23.9]

13. Secondary Outcome: Change in Plasma Brain N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) From Baseline to Weeks 12 and 24
Description: NT-proBNP was assessed at Baseline, Weeks 12 and 24.
Time Frame: Baseline to Weeks 12 and 24
Population: All subjects with data available at Baseline and Weeks 12 and 24.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Treprostinil Injection
Number analyzed (Participants) | 9
pg/mL
  Change from Baseline to Week 12 | -628 [-3854 to -29]
  Change from Baseline to Week 24 | -478 [-1298 to 81.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 24-week study as well as for 4 weeks after completion of the final visit.
Arm/Group | Treprostinil Injection
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Injection (N=13)
Chronic hepatic failure (Hepatobiliary disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (3)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infusion site cellulitis (Infections and infestations) | 1 (1)
Infusion site pain (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Injection (N=13)
Nausea (Gastrointestinal disorders) | 10 (10)
Headache (Nervous system disorders) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 7 (9)
Infusion site pain (General disorders) | 5 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Urinary tract infection (Infections and infestations) | 3 (8)
Infusion site infection (Infections and infestations) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood uric acide increased (Investigations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Device leakage (General disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dyspepsia (General disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion site erythema (General disorders) | 1 (1)
Infusion site vesicles (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.